CLINICAL TRIAL: NCT05375799
Title: Clinical and Electronic Record for Patients With COVID-19 Treated With the Assisted Breathing Helmet - ELMO in Ceará
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Escola de Saúde Pública do Ceará (Other Government)
Responsible Party: Principal Investigator, Marcelo Alcantara Holanda, Superintendent, Escola de Saúde Pública do Ceará
Other Study IDs: 4.833.400
Record Dates: First submitted 2022-05-14; First posted 2022-05-17 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: Acute breathing insufficiency; Continuous Positive Airway Pressure; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 in use of ELMO: This is an observational study, so there are no interventions. Data will be recruited from adult patients diagnosed with COVID-19, described in medical records, by laboratory detection of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) RNA, who used the Assisted Breathing Helmet - ELMO.
  Interventions: Other: Clinical Observation

INTERVENTIONS:
Other: Clinical Observation — This is an observational study, so there are no interventions. Data will be recruited from adult patients diagnosed with COVID-19, described in medical records, by laboratory detection of SARS-CoV-2 RNA, who used the Assisted Breathing Helmet - ELMO.
  All the following predictor variables will be collected: demographic and anthropometric data; clinical characteristics of patients (comorbidities, date of onset of symptoms and initial symptoms, hospital admission, laboratory tests, chest X-ray tests, need for intubation or ICU admission); start date of ELMO use, blood gas analysis before and after the first application of ELMO and data related to its use (number of applications, number of days of therapy, total time of therapy, as well as reasons for the interruption and adverse effects ).

SUMMARY:
Continuous positive airway pressure (CPAP) with a helmet-like interface has been described as a safe strategy, with minimal contamination of the environment, improving the oxygenation of patients with acute respiratory failure (ARF) by COVID-19, avoiding intubation in more than half of the cases. ELMOcpap, developed in Ceará, was a great ally in the treatment of these cases during the pandemic in the state. It is estimated that among public and private services, more than 1.400 ELMOs have been applied to patients with COVID-19. However, the determining factors of the success and failure of its use in the different institutions in which it has been applied are still unknown. Therefore, it is necessary to survey all data associated with the use of the device.

Objectives: 1. To describe the effects of ELMO in the treatment of patients with hypoxemic respiratory failure due to COVID-19 in a database, in a systematic and standardized way, on clinical history, efficacy, safety, modes, duration of use, the occurrence of adverse events and early predictors of failure. 2. Determine the intubation rate of patients with COVID-19 hypoxemic respiratory failure who used the ELMO. 3. Identify the mortality rate of patients with hypoxemic respiratory failure due to COVID-19 who used the ELMO.

Methods: This is a retrospective, multicenter, observational, cohort study of recorded data from patients with COVID-19 hypoxemic respiratory failure who were treated with the ELMO. An online electronic form will be developed with REDCap, where the responsible investigator of each institution will be responsible for filling in the participants' data, ensuring adherence to the protocol and analysis will be carried out of the data of the patients of the participating services of the research that used the ELMO as treatment.

DETAILED DESCRIPTION:
An online electronic form will be developed with REDCap, where the responsible investigator of each institution will be responsible for filling in the participants' data, ensuring adherence to the protocol.

The researchers involved will undergo qualified training and will receive a video, showing step-by-step how REDCap works, so that there are no doubts about the data collection process and to ensure the standardization of the collection protocol.

An explanation of the nature and objectives of the study will be presented to the research subjects, as well as its importance to society, health professionals and researchers.

The investigators will visit the hospital at least five times a week in the morning, afternoon and/or night shifts, for data collection, with monitoring and collection of outcomes being performed daily.

ELIGIBILITY:
Inclusion Criteria:

* Data from adult patients diagnosed with COVID-19 described in medical records by laboratory detection of RNA of SARS-CoV-2, who used the Assisted Breathing Helmet - ELMO, will be recruited.

Exclusion Criteria:

* Illegible medical records or forms or with incomplete data that make it impossible to collect data will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19, confirmed by laboratory detection of SARS-CoV-2 RNA, who used the Assisted Breathing Helmet - ELMO in referral hospitals in Fortaleza, Brazil.
  Data will be collected retrospectively from adult patients admitted to the ICU and wards during the COVID-19 pandemic in Fortaleza.
  An online electronic form will be developed with REDCap, where the responsible investigator of each institution will be responsible for filling in the participants' data, ensuring adherence to the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Risk factors for intubation | up to 60 days
  To evaluate the risk factors for intubation of patients with hypoxemic ARF due to COVID-19 who used the Assisted Breathing Helmet - ELMO.
Risk factors for death | up to 90 days
  To evaluate the risk factors for death of patients with hypoxemic ARF due to COVID-19 who used the Assisted Breathing Helmet - ELMO.

SECONDARY OUTCOMES:
Time to start ELMO therapy | up to 28 days
  Time to start using the Assisted Breathing Helmet - ELMO
Total time of use ELMO therapy | up to 60 days
  Total time of use of the Assisted Breathing Helmet - ELMO
Adverse events of ELMO | up to 60 days
  Adverse events with the use of the Assisted Breathing Helmet - ELMO

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A Holanda, PHD, Principal Investigator — Escola Saude Publica
Locations (1):
- Hospital Leonardo Da Vinci, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The investigators haven't developed a plan for sharing, but would be open to share unidentified data for research or public health purposes.